CLINICAL TRIAL: NCT06262594
Title: Lemborexant Treatment of Insomnia Linked to Epilepsy
Acronym: L'ÉTOILE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: L'ÉTOILE
Record Dates: First submitted 2023-12-21; First posted 2024-02-16 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Epilepsy; Sleep
MeSH Terms: conditions — Epilepsy | interventions — lemborexant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo First (Placebo Comparator): 0mg
  Interventions: Drug: Lemborexant; Drug: Placebo
- Investigational Product First (Active Comparator): 10mg qhs
  Interventions: Drug: Lemborexant; Drug: Placebo

INTERVENTIONS:
Drug: Lemborexant — Drug is administered
  Other Names: Dayvigo
Drug: Placebo — Drug is administered

SUMMARY:
The goal of this clinical trial is to assess whether Lemborexant can improve sleep in patients with epilepsy.

ELIGIBILITY:
Inclusion Criteria:

* Sleep-related focal epilepsy
* Contraception

Exclusion Criteria:

* Changes in antiseizure medication 1 month before study protocol or during study protocol
* Concomitant medications per SUNRISE1
* Individuals with hepatic impairment
* Female participants who are pregnant or breastfeeding
* Individuals with compromised respiratory function
* Individuals with a history of complex sleep-related behaviour
* Individuals with rare hereditary diseases of galactose intolerance such as galactosemia or glucose-galactose malabsorption
* Individuals with a history of dependence or tolerance - abuse, dependence, rebound insomnia
* Individuals with psychiatric disorders with abnormal thinking and behavioural changes, depression, or suicidal ideation
* Individuals with a diagnosis of narcolepsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2024-10-29 (Actual); Primary Completion 2026-04-18 (Estimated); Study Completion 2027-04-18 (Estimated)

PRIMARY OUTCOMES:
WASO | 36 Days
  Wake After Sleep Onset (recorded using PSG)

CONTACTS AND LOCATIONS:
Locations (2):
- Duke University, Durham, North Carolina, United States
- Health Sciences Centre, Winnipeg, Manitoba, Canada